CLINICAL TRIAL: NCT01512030
Title: Prospective Study of Peripherla Neuropathy in Diabetic Type I
Brief Title: Prevalence of Peripheral Neuropathy in Children and Adolescents With Type I Diabetes Mellitus: a Prospective Study
Status: Completed | Type: Observational
Sponsor: Landeskrankenhaus Feldkirch (Other)
Responsible Party: Principal Investigator, Burkhard Simma, Medical Doctor, Professor, Landeskrankenhaus Feldkirch
Other Study IDs: 02
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus Type I; Diabetic Peripheral Neuropathy; Nerve Conduction Study Not Performed
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diabetes mellitus type I is an increasing burden for more and younger children. Therapy should avoid long-term complications as macrovascular diseases and diabetic nephropathy, retinopathy and diabetic neuropathy (DN). There is considerable uncertainty about the prevalence of DN due to a lack of large epidemiological studies and consensus on diagnostic criteria. Nerve conduction velocity studies are regarded as the "gold standard" for investigating neuropathies.

We plan a prospective study by investigating the peripheral nerve conduction velocity in a population of diabetic children. At the same time-points, we will do a neurological examination using the Young Score, a clinical score of peripheral neuropathy [10]. The results obtained will be related to other long-term vascular complications (nephropathy, retinopathy), glycaemic control, duration of diabetes, insulin dose regime, hours of sports/week, and BMI

DETAILED DESCRIPTION:
The number of newly diagnosed patients with diabetes mellitus type I increases every year, with the patients becoming younger. The Austrian Diabetes Incidence Study Group demonstrated a significant and constant increase in the incidence rate from 12.0 to 18.4/100,000 in children and adolescents ≤15 years of age from 1999 to 2007 [7]. So, we are confronted with more and more children and adolescents suffering from complications which determine long-term outcome. Chronic disease and complications have an important impact on quality and expectation of life and on health resources.

Among the long-term complications of diabetes, vascular complications including retinopathy, nephropathy, neuropathy, and macrovascular disease are the most prevalent [2]. The main therapeutic goal is to avoid these complications by early detection of clinical or, even better, subclinical signs. For this reason, the International Society for Pediatric and Adolescent Diabetes (ISPAD) periodically issues Clinical Practice Consensus Guidelines, particularly for screening for vascular complications [2]. With regard to diabetic neuropathy (DN) there is still uncertainty about the time frame, intensity and diagnostic method of choice, despite it is a significant source of morbidity and mortality [3]. Additionally, there is considerable uncertainty about the prevalence of DN due to a lack of large epidemiological studies and consensus on diagnostic criteria [4].

The American Academy of Neurology suggests a combination of objective and symptoms, signs and electrophysiology provides the most accurate diagnosis of distal symmetric polyneuropathy [5]. Nerve conduction studies are considered by many as the "gold standard" for nerve damage and the most consistent indicator of (sub-)clinical neuropathy [6].

So far, several cross-sectional studies have been conducted on nerve conduction velocity in diabetic children. The results in regard of prevalence are largely divergent. We found that 15 out of 39 patients (38.5%) had a pathological nerve conduction velocity. This result neither correlated to a clinical symptom score (Young Score which consist of a Neurological Deficiency Score, NDS and a Neuropathy Symptom Score, NSS) [10], nor to mean HbA1c, patients age, duration of diabetes, body mass index, insulin regime, hours of sports or metabolic testing results.

Only one long-term prospective study addressing the issue of the development of diabetic neuropathy in a juvenile population was done so far [8]. To better understand the long term development of diabetic neuropathy we plan to study the peripheral nerve conduction velocity in a population of diabetic children from our outpatient clinic. At the same time, we will do a neurological examination using the Young Score, a clinical score of peripheral neuropathy [10].

The results obtained will be related to other long-term vascular complications (nephropathy, retinopathy), glycaemic control, duration of diabetes, insulin dose regime, hours of sports/week, and BMI

ELIGIBILITY:
Inclusion Criteria:

* 8 to 18 years suffering from diabetes mellitus type I for more than one year.

Exclusion Criteria:

* Children who are unable to understand informed consent
* Diabetic children with duration of diabetes < 1 year, age <8 or >18
* Insulin < 0.5IE/kg/d
* Blood glucose before examination below 50 or above 350mg/dL
* Children with chronic diseases, handicapped children, children with cancer, chronic renal impairment, or neurological diseases
* Children who are on medications that can produce peripheral neuropathy, i.e antineoplastic drugs

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents 8 to 18 years suffering from diabetes mellitus type I for more than one year.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
What is the long term development of diabetic neuropathy? Is there a significant deterioration or improvement in nerve conduction during the follow up period? | 5-years

SECONDARY OUTCOMES:
Correlation to mean HbA1c | 5 years
mean BMI | 5 years
Blood pressure | 5 years
Retinopathy | 5 years
Nephropathy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Simma, MD, Principal Investigator — Dep. of Pedaitrics Academic Teaching Hospital, Landeskrankenhaus Feldkirch
Locations (1):
- Dep. of Pediatrics, Academic Teaching Hospital, Landeskrankenhaus Feldkirch, Feldkirch, Austria